CLINICAL TRIAL: NCT02916277
Title: Endocan; Can be a New Biomarker in Ventilator-associated Pneumonia?
Brief Title: Endocan in Ventilator-associated Pneumonia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Erzincan University (Other)
Responsible Party: Principal Investigator, ILKE KUPELI, assist. prof., Erzincan University
Other Study IDs: ERZINCAN UNIVERSITY 3
Record Dates: First submitted 2016-09-24; First posted 2016-09-27 (Estimated); Last update posted 2016-09-27 (Estimated); Status verified 2016-09

CONDITIONS: Serial Endocan Measurements

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Days
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: endocan — to look series Endocan level for 5 days in intubated patients

SUMMARY:
In this study; in patients undergoing mechanical ventilation, making the day series Endocan measurements during the first 5 day to look at whether there is a relationship between the levels of VAP with Endocan. This relationship, if any, aimed to investigate whether correlated with clinical and laboratory findings [presence of fever, pathological lung X-ray, the number of white blood cells (WBC), procalcitonin (PCT), C-reactive protein (CRP)] .

ELIGIBILITY:
Inclusion Criteria:

* over 18 age
* Patients whether intubated and connected to a mechanical ventilator

Exclusion Criteria:

* patients intubated due to lung problems such as COPD, asthma, pulmonary embolism , etc.
* Patients with brain tumors
* patients with acute and chronic renal failure
* Patients with hypertension
* Patients with previously diagnosed infection
* Patients with extubated
* patients using antibiotics or corticosteroids before bronchoalveolar lavage fluid samples taken

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients whether intubated and connected to a mechanical ventilator
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2016-08; Primary Completion 2017-02 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
relationship between the level of Endocan and development of VAP | 9 month

SECONDARY OUTCOMES:
correlation with the level of Endocan and clinical and laboratory findings | 9 month

CONTACTS AND LOCATIONS:
Locations (1):
- Erzincan University, Erzincan, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fagon JY, Chastre J, Wolff M, Gervais C, Parer-Aubas S, Stephan F, Similowski T, Mercat A, Diehl JL, Sollet JP, Tenaillon A. Invasive and noninvasive strategies for management of suspected ventilator-associated pneumonia. A randomized trial. Ann Intern Med. 2000 Apr 18;132(8):621-30. doi: 10.7326/0003-4819-132-8-200004180-00004. PMID 10766680
- [Background] Mayhall CG. Ventilator-associated pneumonia or not? Contemporary diagnosis. Emerg Infect Dis. 2001 Mar-Apr;7(2):200-4. doi: 10.3201/eid0702.010209. PMID 11294706
- [Background] Gibot S, Cravoisy A, Levy B, Bene MC, Faure G, Bollaert PE. Soluble triggering receptor expressed on myeloid cells and the diagnosis of pneumonia. N Engl J Med. 2004 Jan 29;350(5):451-8. doi: 10.1056/NEJMoa031544. PMID 14749453
- [Background] Bechard D, Gentina T, Delehedde M, Scherpereel A, Lyon M, Aumercier M, Vazeux R, Richet C, Degand P, Jude B, Janin A, Fernig DG, Tonnel AB, Lassalle P. Endocan is a novel chondroitin sulfate/dermatan sulfate proteoglycan that promotes hepatocyte growth factor/scatter factor mitogenic activity. J Biol Chem. 2001 Dec 21;276(51):48341-9. doi: 10.1074/jbc.M108395200. Epub 2001 Oct 5. PMID 11590178
- [Background] Bechard D, Meignin V, Scherpereel A, Oudin S, Kervoaze G, Bertheau P, Janin A, Tonnel A, Lassalle P. Characterization of the secreted form of endothelial-cell-specific molecule 1 by specific monoclonal antibodies. J Vasc Res. 2000 Sep-Oct;37(5):417-25. doi: 10.1159/000025758. PMID 11025405
- [Result] Luyt CE, Combes A, Reynaud C, Hekimian G, Nieszkowska A, Tonnellier M, Aubry A, Trouillet JL, Bernard M, Chastre J. Usefulness of procalcitonin for the diagnosis of ventilator-associated pneumonia. Intensive Care Med. 2008 Aug;34(8):1434-40. doi: 10.1007/s00134-008-1112-x. Epub 2008 Apr 18. PMID 18421435
- [Result] Linssen CF, Bekers O, Drent M, Jacobs JA. C-reactive protein and procalcitonin concentrations in bronchoalveolar lavage fluid as a predictor of ventilator-associated pneumonia. Ann Clin Biochem. 2008 May;45(Pt 3):293-8. doi: 10.1258/acb.2007.007133. PMID 18482918
- [Result] Flanagan PG, Jackson SK, Findlay G. Diagnosis of gram negative, ventilator associated pneumonia by assaying endotoxin in bronchial lavage fluid. J Clin Pathol. 2001 Feb;54(2):107-10. doi: 10.1136/jcp.54.2.107. PMID 11215277
- [Result] el-Ebiary M, Torres A, Gonzalez J, Martos A, Puig de la Bellacasa J, Ferrer M, Rodriguez-Roisin R. Use of elastin fibre detection in the diagnosis of ventilator associated pneumonia. Thorax. 1995 Jan;50(1):14-7. doi: 10.1136/thx.50.1.14. PMID 7886642
- [Result] Lassalle P, Molet S, Janin A, Heyden JV, Tavernier J, Fiers W, Devos R, Tonnel AB. ESM-1 is a novel human endothelial cell-specific molecule expressed in lung and regulated by cytokines. J Biol Chem. 1996 Aug 23;271(34):20458-64. doi: 10.1074/jbc.271.34.20458. PMID 8702785
- [Result] Tang L, Zhao Y, Wang D, Deng W, Li C, Li Q, Huang S, Shu C. Endocan levels in peripheral blood predict outcomes of acute respiratory distress syndrome. Mediators Inflamm. 2014;2014:625180. doi: 10.1155/2014/625180. Epub 2014 Jul 16. PMID 25132734
- [Derived] Kupeli I, Salcan S, Kuzucu M, Kuyrukluyildiz U. Can endocan be a new biomarker in ventilator-associated pneumonia? Kaohsiung J Med Sci. 2018 Dec;34(12):689-694. doi: 10.1016/j.kjms.2018.07.002. Epub 2018 Aug 9. PMID 30527203